CLINICAL TRIAL: NCT02077192
Title: A Phase 3 Open Label Extension Study of Fostamatinib Disodium in the Treatment of Persistent/Chronic Immune Thrombocytopenic Purpura
Brief Title: Open Label Study of R788 in the Treatment of Persistent/Chronic Immune Thrombocytopenic Purpura (ITP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-935788-049; 2013-005454-30 (EudraCT Number)
Record Dates: First submitted 2014-02-27; First posted 2014-03-04 (Estimated); Results first posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Immune Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — fostamatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fostamatinib Disodium (Experimental): Fostamatinib Disodium tablet 100 mg or 150 mg by mouth twice a day
  Interventions: Drug: Fostamatinib Disodium

INTERVENTIONS:
Drug: Fostamatinib Disodium — Fostamatinib Disodium tablet 100 mg or 150 mg by mouth twice a day
  Other Names: R935788; R788; Fostamatinib

SUMMARY:
The primary objective of this study was to assess the long term safety of fostamatinib in subjects with persistent/chronic ITP

ELIGIBILITY:
Inclusion Criteria:

* Completed week 24 evaluation of Study C935788-047 or Study C935788-048 or discontinued early due to lack of response.
* Able and willing to give written informed consent

Exclusion Criteria:

* Discontinued participation in Study C935788-047 or Study C935788-048 for any reason other than lack of response
* Poorly controlled hypertension during Study C935788-047 or Study C935788-048
* Significant infection, an acute infection such as influenza, or known inflammatory process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2014-10; Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rigel Pharmaceuticals, Inc., Study Director — Rigel Pharmaceuticals,Inc.
Locations (55):
- United States (9):
  - Arizona Oncology Associates, Tucson, Arizona
  - Bleeding & Clotting Disorders Institute, Peoria, Illinois
  - Horizon Oncology Research, Inc, Lafayette, Indiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Weill Cornell Medical College/New York Presbyterian Hospital, New York, New York
  - Weill Cornell Medicine, New York, New York
  - East Carolina University, Brody School of Medicine, Greenville, North Carolina
  - W.G. "Bill" Hefner VA Medical Center, Salisbury, North Carolina
  - Signal Point Clinical Research Center LLC, Middletown, Ohio
- Australia (7):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Launceston General Hospital, Launceston, Tasmania
  - The Alfred, Melbourne, Victoria
  - Perth Blood Institute, Nedlands, Western Australia
- Hanusch-Krankenhaus Wiener Gebietskrankenkasse, Vienna, Austria
- Bulgaria (4):
  - Specialized Hospital for Active Treatment of Hematology Diseases, EAD, Sofia, Department of Chemotherapy, Hemotherapy and Blood Inherited Diseases to Clinic of Clinical Hematology;, Sofia, BG
  - UMHAT Dr. Georgi Stranski, EAD, Pleven, Clinic of Hematology, Pleven
  - UMHAT Aleksandrovska, EAD, Sofia
  - MHAT Hristo Botev, AD, Vratsa, First Internal Department, Vratsa
- Canada (2):
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - St. Michael's Hospital, Toronto, Ontario
- Czechia (2):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Ostrava, Ostrava-Poruba
- Herlev Hospital, Herlev, DK, Denmark
- Pecsi Tudomanyegyetem Klinikai Kozpont, I. sz. Belgyogyaszati Klinika, Pécs, Hungary
- Italy (2):
  - Istituto di Ematologia "Lorenzo e Ariosto Seràgnoli", Bologna, BO
  - Azienda Ospedaliero-Universitaria "Santa Maria della Misericordia" - Clinica Ematologica, Udine
- HAGA ziekenhuis, The Hague, NL, Netherlands
- Norway (2):
  - Haukeland universitetssykehus, Helse Bergen HF, Bergen
  - Sykehuset Østfold Kalnes, Grålum
- Poland (8):
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 we Wrocrlaw, Wroclaw, Dolnoslaski
  - Wojewodzki Szpital Specjalistyczny im. J. Korczaka, Słupsk, PO
  - Lkinika Hematologii I Transplantologii Uniwersyteckie Centrum Kliniczne, Gdansk
  - SPZOZ Szpital Uniwersytecki w Krakowie Pracownia Separacji Krwinek i Bank Komórek Krwiotwórczych Klinika Hematologii, Krakow
  - Wojewódzki Szpital Specjalistyczny im. M. Kopernika w Łodzi, Lodz
  - Specjalistyczny Gabinet Lekarski, Lublin
  - Szpital Wojewodzki w Opolu, Opole
  - Instytut Hematologii I Transfuzjologii, Warsaw
- Spitalul Clinic Colentina, Hematologie, Bucharest, Romania
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitari i Politécnic La Fe de Valencia, Valencia
- United Kingdom (11):
  - Colchester General Hospital, Colchester, Essex
  - Royal Victoria Infirmary, Newcastle upon Tyne, UK
  - Kent & Canterbury Hospital, Canterbury
  - James Paget University Hospital, Great Yarmouth
  - St. James's Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Royal Liverpool University Hospital, Liverpool
  - Imperial College Healthcare NHS Trust, London
  - University College Hospital, London
  - Cancer and Haematology Centre, Oxford
  - University Hospital of North Midlands NHS Trust, Royal Stoke University Hospital, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cooper N, Altomare I, Thomas MR, Nicolson PLR, Watson SP, Markovtsov V, Todd LK, Masuda E, Bussel JB. Assessment of thrombotic risk during long-term treatment of immune thrombocytopenia with fostamatinib. Ther Adv Hematol. 2021 Apr 30;12:20406207211010875. doi: 10.1177/20406207211010875. eCollection 2021. PMID 33995988

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 124 subjects were screened from studies C788-047/ C788-048 for this extension study. Out of which, 123 subjects were enrolled and treated with study drug.
Groups:
- Fostamatinib Disodium: Fostamatinib was self-administered twice daily (bid) by orally, once in the morning and once in the evening for up to 5 years or until commercial availability of fostamatinib for all subjects, whichever occurred first, in 2 dosage strengths: 100 milligram (mg) and 150 mg.
Period: Overall Study
Arm/Group | Fostamatinib Disodium
Started | 123
Completed | 29
Not Completed | 94

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are analyzed with treated population data analysis set which was defined as all enrolled and treated subjects.
Groups:
- Overall Study: Baseline characteristics are analyzed with treated population data analysis set which was defined as all enrolled and treated subjects.
Arm/Group | Overall Study
Number analyzed (Participants) | 123
Age, Continuous [Median (Full Range); unit: years] | 52.0 [20 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 121
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 113
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Romania | 1
  Hungary | 2
  United States | 17
  Czechia | 10
  United Kingdom | 18
  Spain | 4
  Canada | 4
  Austria | 1
  Netherlands | 1
  Norway | 2
  Poland | 34
  Denmark | 1
  Italy | 6
  Bulgaria | 12
  Australia | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Achieved Platelet Count of at Least 50,000/µL Within 12 Weeks of Beginning Treatment up to 12 Months (Fostamatinib in 047/048 or 049):Version 1
Description: Percentage of subjects who achieved platelet count of at least 50,000/µL within 12 Weeks of beginning treatment up to 12 months was analyzed among all subjects who received active treatment in one of the prior studies (C788-047 or C788-048), in the current extension study (C788-049), or in both prior and current studies. Treated Population was defined as all enrolled and treated subjects.
Time Frame: Up to 12 months
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Fostamatinib Disodium
Number analyzed (Participants) | 123
Percentage of Subjects | 15.4 [9.6 to 23.1]

2. Primary Outcome: Percentage of Subjects Who Achieved Platelet Count of at Least 50,000/µL Within 12 Weeks of Beginning Treatment up to 12 Months (Placebo in 047/048 and Fostamatinib 049): Version 2
Description: A within-subject, between-study comparison of platelet counts for subjects who were previously treated with placebo in one of the prior studies (C788-047 or C788-048) was prospectively defined in the protocol (version 2). Achievement of platelet response by 12 weeks and maintenance of platelet response for 12 weeks was analyzed among subjects who had been randomized to placebo in one of the prior studies (C788-047 or C788-048). Treated Population was defined as all enrolled and treated subjects.
Time Frame: Up to 12 months
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Fostamatinib Disodium
Number analyzed (Participants) | 123
Percentage of Subjects | 2.3 [0.1 to 12.0]

3. Secondary Outcome: Duration of Platelet Response Based on Platelet Count and Rescue Medication
Description: The duration of platelet response was defined as the time from when the subject first achieved a platelet count of at least 50,000/µL, until the first of 2 visits with platelet counts < 50,000/µL that were at least 4 weeks apart without an intervening visit with a platelet count less than equal to (<=) 50,000/µL unrelated to rescue therapy. Duration of platelet response was analyzed using the Kaplan-Meier method. Treated Population was defined as all enrolled and treated subjects. Here, a number of subjects analyzed included all subjects evaluable for this endpoint.
Time Frame: Up to 12 months
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Fostamatinib Disodium: Fostamatinib Disodium tablet 100 mg by mouth twice a day or 150 mg by mouth twice a day
Arm/Group | Fostamatinib Disodium
Number analyzed (Participants) | 57
Days | 127.0 [71.0 to 483.0]

4. Secondary Outcome: Percentage of Subjects in Whom a Reduction in the Dose of Concomitant ITP Therapy Can be Achieved While Maintaining an Adequate Platelet Count
Description: The percentage of subjects in whom a reduction in the dose of concomitant ITP therapy could be achieved while maintaining an adequate platelet count, the reduction event was clarified to apply only to reductions in the dose of concomitant ITP therapy occurring within a period of platelet response and the reduction event was not be prompted by an adverse event.
Time Frame: Up to 12 months
Population: insufficient of number participants with events to perform the analysis
Arm/Group | Fostamatinib Disodium
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 62 months
Arm/Group | Fostamatinib Disodium
All-Cause Mortality (participants affected / at risk) | 4/123
Serious Adverse Events (participants affected / at risk) | 34/123
Other Adverse Events (participants affected / at risk) | 98/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fostamatinib Disodium (N=123)
Aortic stenosis (Vascular disorders) | 1
Chest pain (General disorders) | 1
Mucosal haemorrhage (General disorders) | 1
Pyrexia (General disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Transaminases increased (Investigations) | 2
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Headache (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Hematochezia (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Sepsis (Infections and infestations) | 2
Cellulitis staphylococcal (Infections and infestations) | 1
Endocarditis bacterial (Infections and infestations) | 1
Erythema induratum (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Mastoiditis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Viral Infection (Infections and infestations) | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fostamatinib Disodium (N=123)
Hypertension (Vascular disorders) | 22 (32)
Contusion (Injury, poisoning and procedural complications) | 12 (23)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (19)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 (27)
Headache (Nervous system disorders) | 15 (26)
Fatigue (General disorders) | 10 (11)
Pyrexia (General disorders) | 7 (13)
Diarrhoea (Gastrointestinal disorders) | 36 (62)
Vomiting (Gastrointestinal disorders) | 11 (14)
Petechiae (Skin and subcutaneous tissue disorders) | 19 (31)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8)
Nasopharyngitis (Infections and infestations) | 9 (14)
Upper respiratory tract infection (Infections and infestations) | 14 (20)
Dizziness (Nervous system disorders) | 13 (13)
Nausea (Gastrointestinal disorders) | 11 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (12)
Edema peripheral (General disorders) | 7 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT02077192/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-27): https://cdn.clinicaltrials.gov/large-docs/92/NCT02077192/SAP_001.pdf